CLINICAL TRIAL: NCT01850433
Title: Internet-based Cognitive Behavior Therapy for Body Dysmorphic Disorder: A Pilot Study
Brief Title: Internet Cognitive Behavior Therapy (CBT) for Body Dysmorphic Disorder (BDD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Christian Rück, Associate professor, M.D., Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BDD-P
Record Dates: First submitted 2013-05-07; First posted 2013-05-09 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Body Dysmorhpic Disorder
Keywords: BDD; CBT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Internet CBT (Experimental)
  Interventions: Behavioral: Internet based CBT for body dysmorphic disorder

INTERVENTIONS:
Behavioral: Internet based CBT for body dysmorphic disorder

SUMMARY:
The primary aim is to develop, and test the feasibility, of a novel and protocol-based cognitive behaviour therapy (CBT) treatment for body dysmorphic disorder (BDD) administered via the Internet.

ELIGIBILITY:
Inclusion Criteria:

* outpatients
* male or female

  -≥ 18 years
* currently living in Stockholm county
* primary diagnosis of BDD according to the DSM-IV-TR
* signed informed consent
* regular access to a computer with Internet access and skills to use the web.

Exclusion Criteria:

* psychotropic medication changes within two months prior to the treatment
* completed CBT for BDD within the last 12 months
* BDD-YBOCS < 12 at psychiatrist visit
* other primary axis I diagnosis
* current substance dependence
* lifetime bipolar disorder or psychosis
* suicidal ideation
* Axis II diagnosis that could jeopardize treatment participation
* other current psychological treatment that could affect BDD symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Body dysmorphic disorder symptoms | Measured after 12 weeks of treatment, and after 3 months after treatment

SECONDARY OUTCOMES:
Functioning and life satisfaction | After 12 weeks of treatment, and 3 months after treatment
Depressive symptoms | After 12 weeks of treatment, and 3 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christian Rück, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- M46 Huddinge sjukhus, Internetpsykiatrienheten/mottagningen för tvångssyndrom, Stockholm, Sweden

REFERENCES:
- [Result] Enander J, Ivanov VZ, Andersson E, Mataix-Cols D, Ljotsson B, Ruck C. Therapist-guided, Internet-based cognitive-behavioural therapy for body dysmorphic disorder (BDD-NET): a feasibility study. BMJ Open. 2014 Sep 25;4(9):e005923. doi: 10.1136/bmjopen-2014-005923. PMID 25256187
- See also: Results BMJ Open paper — http://bmjopen.bmj.com/content/4/9/e005923